CLINICAL TRIAL: NCT03911024
Title: Development and Piloting of a Just-in-Time, Personalized HIV Prevention Intervention for Youth Experiencing Homelessness (YEH) and Unstable Housing (Study Alias: HIV Prevention Messaging Intervention for YEH)
Brief Title: Development and Piloting of a Just-in-Time, Personalized HIV Prevention Intervention for Youth Experiencing Homelessness and Unstable Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Diane Santa Maria, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SN-18-0501
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Behavior, Risk
Keywords: HIV prevention; homeless
MeSH Terms: conditions — Risk-Taking | interventions — Health Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV (Active Comparator)
  Interventions: Behavioral: HIV
- General Health (Placebo Comparator)
  Interventions: Behavioral: General health

INTERVENTIONS:
Behavioral: HIV — At the completion of each EMA, participants in the intervention group (n=50) will receive messages that address:1) unsafe sexual behaviors, 2) alcohol/drug use, 3) PrEP interest, and 4) HIV testing. In addition, participants will have access to a button in the app that will link them to resources when/if they are the victim of sexual assault. Finally, intervention arm youth will be asked to set a behavioral goal related to HIV prevention during this session. Those goals will include increasing condom use, PrEP use, non-occupational post-exposure prophylaxis (nPEP) use, reducing number of sexual partners, not having sex with using drugs or drinking alcohol, avoiding IV drug use, getting testing for HIV, and testing and treating sexually transmitted infections (STIs) as needed
  Arms: HIV
Behavioral: General health — Participants in the attention control condition (n=50) will answer the same EMA items as the Intervention group. However, the intervention messages will contain content related to nutrition, physical activity, sleep hygiene, and tobacco use. Finally, control arm youth will be asked to set a behavioral goal related to general health during this session.Those goals will include getting 7+ hours of sleep, eating >= 5 servings of fruits or vegetables, not using tobacco products, exercising at least 60 minutes.
  Arms: General Health

SUMMARY:
The purpose of this study is develop and pilot test a personalized HIV intervention with youth experiencing homelessness by creating and field testing prevention messages that address real-time predictors (e.g., sexual urge, use to use drugs, and substance use) of HIV risk behaviors,to evaluate the feasibility and acceptability of the intervention and to evaluate the intervention outcome effects on HIV risk behaviors (e.g., condomless sex, number of sexual partners, pre-exposure prophylaxis(PrEP) awareness, substance use during sex,Intravenous(IV)drug use)

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* HIV high risk: IV drug user or sexually active youth (sex in the past 3 months) who reports at least one of the following: condomless sex, concurrent sexual partners within 2 weeks,sex with a partner of unknown HIV status, or a bacterial STI in the last 6 months.
* Homelessness: staying on the streets or in a place not meant for human habitation, a shelter,hotel/motel, or some place they cannot stay for more than 30 days

Exclusion Criteria:

* Below 6th grade reading level:determined by the Rapid Estimate of Adult Literacy in Medicine Short Form (REALM)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by number recruited | baseline
  Number recruited is number of eligible youth minus number who refuse to participate.
Feasibility as assessed by number of participants who complete the study | 6 weeks
Feasibility as assessed by number of staff hours required | 6 weeks
Feasibility as assessed by number of participants who damage or lose phones | 6 weeks
Acceptability as assessed by score on the System Usability Scale (SUS) | 6 weeks
  The System Usability Scale (SUS) consists of 10 items on a 5-point (0-4) Likert scale and is designed to assess acceptability of a product. Overall score ranges from 0 to 100, with higher scores indicating greater acceptability.
Acceptability as assessed by score on the Mobile App Rating Scale (MARS) | 6 weeks
  The Mobile App Rating Scale (MARS) consists of 23 items on a 5-point (1-5) scale is designed to score apps on the criteria of engagement, functionality, aesthetics, and information quality (sub-scales). Total score is determined by calculating the mean of each sub-scale and an overall mean score. High mean scores indicate a higher quality app.
Number of participants who complete greater than 80% of the Ecological Momentary Assessments (EMAs) | 6 weeks
Number of participants who read greater than 80% of Just-In-Time Adaptive Intervention (JITAI) messages | 6 weeks
Effect on HIV risk behaviors as assessed by number of participants who use condoms | 6 weeks
Effect on HIV risk as assessed by number who use substances before sex | 6 weeks
Effect on HIV risk as assessed by number of participants who have pre-exposure prophylaxis (PrEP) interest | 6 weeks
Effect on HIV risk as assessed by number of participants who undergo HIV or sexually transmitted infection (STI) testing | 6 weeks
Effect on HIV risk as assessed by number of sexual partners | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diane Santa Maria, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santa Maria D, Padhye N, Businelle M, Yang Y, Jones J, Sims A, Lightfoot M. Efficacy of a Just-in-Time Adaptive Intervention to Promote HIV Risk Reduction Behaviors Among Young Adults Experiencing Homelessness: Pilot Randomized Controlled Trial. J Med Internet Res. 2021 Jul 6;23(7):e26704. doi: 10.2196/26704. PMID 34255679